CLINICAL TRIAL: NCT03853239
Title: A Randomised, Crossover Comparison of Nasal Ventilation vs Face Mask in Anesthetised Adults
Brief Title: Nasal Ventilation vs Face Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: nasal ventilation vs face mask
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Nasotracheal Intubation
Keywords: face mask; nasal ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face mask crossover nasal ventilation (Active Comparator)
  Interventions: Procedure: face mask ventilation crossover nasal ventilation
- nasal ventilation crossover face mask (Active Comparator)
  Interventions: Procedure: nasal ventilation crossover face mask ventilation

INTERVENTIONS:
Procedure: face mask ventilation crossover nasal ventilation — Group A was first ventilated through the face mask, and the tidal volume was measured under pressure-controlled mode (10, 15, 20 cm H2O) ;Switched to volume-controlled (6,8,10ml/kg predicted body weight)mode, the actual tidal volume was recorded, and the air leakage was calculated. Then, put a nasal RAE tube in one side of the nostril, inflate the cuff, make the catheter in a natural position after inflation, clip the other side of the nostril, close the lip with tape, connect the breathing circuit, record the actual tidal volume; measure the expired tidal volume during pressure-controlled ventilation (10, 15, 20 cm H2O).Subject will start with one technique and then cross over to the other technique.
  Arms: face mask crossover nasal ventilation
Procedure: nasal ventilation crossover face mask ventilation — Group B first placed a nasal RAE tube in one side of the nostril, the cuff was inflated, the catheter was in a natural position after inflation, the other side of the nostril was clamped, the lip was closed with tape, the breathing circuit was connected, and the amount of tidal volume was measured under pressure-controlled mode ( 10,15,20cm H2O) ; switch to volume-controlled ventilation mode (6,8,10ml/kg predicted body weight), record the actual tidal volume; pull out the tracheal tube, perform mask ventilation, record the actual tidal volume and tidal volume under volume-controlled mode(6,8,10ml/kg predicted body weight) and pressure-controlled mode (10, 15, 20 cm H2O) , respectively.Subject will start with one technique and then cross over to the other technique.
  Arms: nasal ventilation crossover face mask

SUMMARY:
Nasotracheal intubation(NTI) is commonly used in operations of the mouth, pharynx, larynx and also the neck. While these patients showed higher rates of difficult laryngoscopy. Therefore, duration of apnoea is prolonged and re-oxygenation is inevitable.Mask ventilation is the most fundamental technique in maintaining oxygenation, even when endotracheal intubation is failed. However, the most common complication of NTI is epistaxis, removing the nasotracheal tube could make mask ventilation extremely difficult.So the investigatorsbelieve the ideal approach is ventilation through original nasotracheal tube.Several techniques of supraglottic ventilations through endotracheal tubes have been reported.It remains uncertain whether supraglottic ventilation through inflated nasal RAE endotracheal tube has similar efficiency as mask ventilation after general anesthesia induction. Based on previous clinical experience, the investigators hypothesised that ventilations through inflated nasal RAE endotracheal tube and through facemask were comparable in terms of tidal volume and airway pressure in anesthetized, apnoeic adults.

Forty patients were randomly assigned (sealed envelope method) to face mask（Group A，n=20）or nasal ventilation(Group B，n=20), For A: face mask ventilation followed by nasal ventilation and for B:nasal ventilation followed by face mask ventilation.Measure the tidal volume and air leakage of face mask and nasal ventilation during pressure-controlled ventilation mode and volume-controlled mode, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years old
* ASA physical status I and II
* Requiring general anesthesia with nasal intubation

Exclusion Criteria:

* Respiratory disease，cardiovascular disease, cerebral vascular disease
* Anticipated Difficult Mask Ventilation(Age>55 years old, obesity,bearded,edentulous,a history of snoring)
* The need for emergency surgery
* Contraindications to nasal intubation
* Pregnancy
* Gastric-esophageal reflex or a full stomach

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in expired tidal volume of each technique under pressure-controlled mode | 3 breaths of expired tidal volume for each technique
Difference in air leakage of each technique under volume-controlled mode | 3 breaths of air leakage for each technique

SECONDARY OUTCOMES:
number of participants with Oxygen Saturation- Reading Below 95% | intraoperative duration of each ventilation technique
peak inspiratory pressure | intraoperative duration of each ventilation technique
end tidal CO2 partial pressure Reading- Median | intraoperative duration of each ventilation technique
hemodynamic changes | intraoperative duration of each ventilation technique

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital,Affililated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China